CLINICAL TRIAL: NCT03823690
Title: EUS-guided Balloon-occluded Gastrojejunostomy Bypass (EPASS) Versus Uncovered Duodenal Stent for Unresectable Malignant Gastric Outlet Obstruction.
Brief Title: EPASS Versus Uncovered Duodenal Stent for Unresectable Malignant Gastric Outlet Obstruction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE-2018.335
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Intervention Model Description: The patients would be randomized to either EUS-guided balloon-occluded gastrojejunostomy bypass (EPASS) or uncovered duodenal stent after cannulation of the obstruction site is achieved with the guide-wire.
Who Masked: Participant
Masking Description: Recruited patients would not be informed of the type of treatment that was received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided gastrojejunostomy (Active Comparator): The procedures would be performed under conscious sedation or monitored anesthesia by a therapeutic gastroscope. The endoscope would be used to reach the site of obstruction. The stricture would be cannulated with a 0.025" or 0.035" guide-wire. The double balloon occluder would then be inserted on guidewire beyond the duodenal-jejunal flexure and the two balloons of the occluder would be inflated.
  A segment of duodenum/jejunum would then be occluded and saline would be injected. A linear echoendoscope would then be inserted into the stomach to guide insertion of the gastrojejunostomy stent.
  Interventions: Device: EUS-guided gastrojejunstomy
- Pyloro-duodenal stent (Active Comparator): The uncovered DS used in this study is Wallflex (Boston, Natick, MA, USA), made of nitinol wire, with a diameter of 22mm and length of 6, 9, 12cm. This stent is a braided stent with high axial force, good flexibility and conformability.
  Interventions: Device: The pyloro-duodenal stent

INTERVENTIONS:
Device: EUS-guided gastrojejunstomy — As listed in the arms description
  Other Names: EPASS
  Arms: EUS-guided gastrojejunostomy
Device: The pyloro-duodenal stent — As listed in the arms description
  Other Names: DS
  Arms: Pyloro-duodenal stent

SUMMARY:
Surgical gastrojejunostomy is the conventional treatment for palliating patients suffering from of inoperable malignant gastric outlet obstruction (GOO). Although, the procedure is associated with a high success and low re-intervention rates, there is a risk of morbidities (10% - 16%) and mortalities (7%). The placement of a pyloro-duodenal self-expandable metallic stent (SEMS) is an alternative to surgery for the palliating these patients. As compared to surgery, the procedure is associated with shorter hospital stay, reduced morbidities and cost. However, the clinical efficacy of SEMS is limited by several problems. In uncovered SEMS, the long-term patency is reduced by tumor ingrowth leading to subsequent re-stenosis. In covered SEMS, stent migration occurs at a frequency of 14-25% and it is a major obstacle to stent patency. As a result, randomized trials comparing uncovered stents and partially or fully covered stents in patients with malignant GOO have reported comparable stent patency between the two types of stents.

Recently, the creation of a gastrojejunostomy under EUS (EUS-GJ) guidance using lumen-apposing stents has been described. The procedure was associated with a technical success rate of around 90% and clinical success of 85% to 100%. The procedure holds the potential to create a gastrojejunostomy without surgery. Furthermore, there is a low risk of tumor ingrowth and stent migration, thus improving the stent patency and reducing the need of re-intervention. We have previously published a novel method of creating EUS-GJ with the use of a double balloon occluder (EPASS). The device provides a stable condition for performance of EUS-GJ and improves the safety of the procedure. However, there is limited data on how EPASS compares to endoscopic stenting. The aim of the current study is thus to compare EPASS and DS under a randomized setting.

DETAILED DESCRIPTION:
In recent years, SEMSs have provided an attractive alternative to surgery for palliation of malignant gastric outlet obstruction. Several studies have assessed the clinical and technical success rates of pyloro-duodenal SEMS for malignant gastroduodenal obstruction. Technical success rates of 90% to 100% and clinical success of 80% to 95% was achieved.The procedure was associated with quicker recovery and reduced morbidities as compared to surgical gastrojeunostomies. However, the long-term patency of uncovered SEMS is limited by the risk of tumor ingrowth that would lead to subsequent re-stenosis of the stents requiring re-intervention. Thus to palliate malignant gastric outlet obstruction, surgical gastrojejunostomy is preferred in patients that are at good risk for surgery with prolonged life expectancy whilst insertion of pyloro-duodenal SEMS is preferred in patients that are associated with high-risk for surgery and short life expectancy.

In lieu of the above reasons, it would be the ideal situation if a gastrojejunostomy could be created endoscopically without surgery. The procedure could potentially avoid the risk of morbidities and mortalities associated with surgery whilst enjoying the superior patency associated with a gastrojejunostomy. However, a number of hurdles need to be overcome for safe creation of an anastomosis endoscopically. Firstly, the collapsed bowel (duodenum or jejunum) needs to be easily identified from the stomach. Secondly, a reliable method of creating an anastomosis needs to be available. Lastly, a device for maintaining the anastomosis between two non-adherent organs is required.

The use of EUS as a platform to create a gastrojejunostomy endoscopically may theoretically tackle all of the above hurdles. The device could be used in the stomach to visualize the adjacent duodenum or jejunum for anastomosis. A 19-gauge needle could be used to puncture the adjacent bowel for passage of a guide-wire to connect the two non-adherent organs. Thereafter, a SEMS could be placed between the two organs for creation and maintenance of the anastomosis.

Initial results of EUS-guided gastrojejunostomies from two studies have become available. Khashab et al reported EUS-GJ in 10 patients. Technical success was achieved in 9 patients (90%). Clinical success with resumption of solid oral intake was achieved in all 9 patients (100%), who underwent successful EUS-GE. 8 patients were able to tolerate almost a normal diet and/or full diet, and 1 patient tolerated a soft diet. There were no procedure-related adverse events. Mean procedure time was 96 minutes (range 45-152 minutes), and mean length of hospital stay was 2.2 days. In another multicenter study, 26 patients received EUS-GJ. Technical success was achieved in 24 patients (92 %). Clinical success was achieved in 22 patients (85 %). Of the 4 patients in whom clinical success was not achieved, 2 had persistent nausea and vomiting despite a patent EUS-GJ and required enteral feeding for nutrition, 1 died before the initiation of an oral diet, and 1 underwent surgery for suspected perforation. Adverse events, including peritonitis, bleeding, and surgery, occurred in 3 patients (11.5 %). In both of these studies, the AXIOS stent was used for creation of the anastomosis (Boston Scientific, Natick, MA, USA).

However, a common technical problem exists in both of these series. The target duodenum or jejunum needed for creation of a GJ is collapsed and it is difficult to identify the target organ by EUS from the stomach. Furthermore, the insertion of the stent for creation of the anastomosis may be difficult with a collapsed bowel and this may result in catastrophic outcomes. Our group has overcome this problem with a novel device - the double balloon occluder. The device comprises of two balloons that could occlude a segment of bowel. Saline could then be injected in to the occluded segment resulting in distension of the bowel and making it possible to be targeted by EUS from the stomach.

Our group has published the results of using the double balloon occluder in conjunction with the AXIOS stent for creation of a GJ in 20 patients (Endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy bypass - EPASS). The technical success rate was 90% (18/20). The median intubation time from the double-balloon tube intubation to stent placement was 25.5 min (range 10-39 min). Post-treatment gastric outlet obstruction scoring system (GOOSS) score improved in all 18 cases in which EPASS was successfully performed. The mean post-GOOSS score was significantly higher than the pre-GOOSS score (0.6±0.75 vs 2.94±0.23, p<0.001). None of the patients with successful placement of the stent suffered from adverse events or recurrent obstruction.

The outcomes of EUS-GJ were recently compared with that of conventional procedures for management of malignant GOO. In a retrospective study, EUS-GJ was compared with DS. 30 patients received EUS-GJ and 60 patients DS. The technical success rates were similar between the two groups (96.7% vs. 86.7%, P=0.07). Clinical success was also similar between the two groups (70.0% vs. 86.7%, P=0.08). The re-intervention rate was significantly higher in the ES group (43.3% vs. 3.4%, P<0.001), whilst adverse events were comparable (13.3% vs 18.3%, P = 0.549). On multivariate analysis, DS was independently associated with need for re-intervention (OR 25.7, p=0.004). In another study, EUS-GJ (25 patients) was compared with laparoscopic gastrojejunostomy (29 patients) 20. Technical success was comparable (88% vs 100%, P = 0.11). Clinical success was similar (84% vs 90%, P = 0.11). Average post-procedure length of stay was 9.4 days in the EUS-GJ group and 8.9 days in the Lap-GJ group (P = 0.75). Adverse events were significantly more the lap-GJ group (41% vs 12%, P = 0.03).

Thus, based on the above results, EUS-GJ may be associated with improved outcomes as compared with conventional procedures for management of malignant GOO. Hence, the aim of the current study is to compare the efficacies of EPASS versus uncovered pyloro-duodenal stents (DS) in unresectable malignant gastric outlet obstruction in a randomized setting.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients ≥ 18 years old
* Confirmed unresectable distal gastric or duodenal or pancreatico-biliary malignancies
* Suffering from gastric outlet obstruction with a gastric outlet obstruction score of ≤ 1
* Performance status ECOG ≤3

Exclusion Criteria:

* Prior metallic stent placement
* Severe comorbidities precluding the endoscopic procedure (such as cardiopulmonary disease, sepsis, or a bleeding disorder)
* Life expectancy of less than 1 month
* History of gastric surgery
* Linitus plastic
* Multiple-level bowel obstruction confirmed on radiographic studies such as small bowel series or abdominal computed tomography
* Coagulation disorders
* Pregnancy
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Re-intervention rate | 6 months
  The percentage of patients requiring additional endoscopic intervention due to stent dysfunction.

SECONDARY OUTCOMES:
Technical success rate | 1 day
  The successful placement of a stent across the site of obstruction, as confirmed by endoscopy or fluoroscopy.
Clinical success rate | 3 days
  Clinical success if measured by the improvement of at least 1 point in the gastric outlet obstruction score within 3 days after stent insertion.
Stent dysfunction rate | 6 months
  Stent dysfunction is defined as the restenosis of the stent due to tumor ingrowth or overgrowth, stent migration, or fracture.
Duration of stent patency | 6 months
  Calculated from the time of stent placement to the time of stent dysfunction.
Adverse events rate | 6 months
  Graded according to the lexicon of endoscopic adverse events
Mortality | 6 months
  Death from any cause
Gastric outlet obstruction scores (GOOS) | 6 months
  Scoring system for food intake. Range of score is 0 -3 with 3 being the highest and indicating tolerating full diet
Quality of life assessment scores | 6 months
  EORTC QLQ-C30. This questionnaire is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of 5 multiitem scales (physical, role, social, emotional and cognitive functioning) and 9 single items (pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life assessment scores | 6 months
  EORTC STO-22 modules. This the gastric cancer module to the QLQ-C30 questionnaire. The questionnaire is composed of 5 multiitem scales (dysphagia, pain, reflux, eating, anxiety) and 4 single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Teoh AYB, Lakhtakia S, Tarantino I, Perez-Miranda M, Kunda R, Maluf-Filho F, Dhir V, Basha J, Chan SM, Ligresti D, Ma MTW, de la Serna-Higuera C, Yip HC, Ng EKW, Chiu PWY, Itoi T. Endoscopic ultrasonography-guided gastroenterostomy versus uncovered duodenal metal stenting for unresectable malignant gastric outlet obstruction (DRA-GOO): a multicentre randomised controlled trial. Lancet Gastroenterol Hepatol. 2025 Jun;10(6):e8-e16. doi: 10.1016/S2468-1253(25)00136-0. PMID 40347959
- [Derived] Teoh AYB, Lakhtakia S, Tarantino I, Perez-Miranda M, Kunda R, Maluf-Filho F, Dhir V, Basha J, Chan SM, Ligresti D, Ma MTW, de la Serna-Higuera C, Yip HC, Ng EKW, Chiu PWY, Itoi T. Endoscopic ultrasonography-guided gastroenterostomy versus uncovered duodenal metal stenting for unresectable malignant gastric outlet obstruction (DRA-GOO): a multicentre randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Feb;9(2):124-132. doi: 10.1016/S2468-1253(23)00242-X. Epub 2023 Dec 4. PMID 38061378